CLINICAL TRIAL: NCT00841633
Title: Induced Hypertension for Delayed Cerebral Ischaemia After Aneurysmal Subarachnoid Haemorrhage:a Feasibility Study
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Our RCT recently started. The RCT is similar to the feasibility trial, so it was terminated to avoid 2 trials running simultaniously.
Sponsor: UMC Utrecht (Other)
Collaborators: Netherlands Organisation for Scientific Research (Other Government)
Responsible Party: Principal Investigator, A.J.C. Slooter, dr. A.J.C. Slooter, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-137
Record Dates: First submitted 2008-10-10; First posted 2009-02-11 (Estimated); Last update posted 2011-10-12 (Estimated); Status verified 2011-10

CONDITIONS: Cerebral Ischemia; Subarachnoid Hemorrhage
Keywords: subarachnoid hemorrhage; ischemia; vasospasm; CT; perfusion; induced hypertension; delayed cerebral ischemia
MeSH Terms: conditions — Brain Ischemia; Subarachnoid Hemorrhage; Ischemia | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): No induced hypertension (reference group)
- 2 (Experimental): Induced hypertension with a MAP of 30 mmHg above the average MAP on the previous day; during 24-36 hours, until a perfusion CT scan has been performed
  Interventions: Drug: Induced hypertension with norepinephrine

INTERVENTIONS:
Drug: Induced hypertension with norepinephrine — Hypertension will be induced with norepinephrine. Administration of norepinephrine results in vasoconstriction, leading to an increase in blood pressure. The normal blood pressure of the patient will be calculated as the average MAP of the day before the start of the study. To achieve the intended hypertension (30 mmHg above the normal MAP for patients allocated to index group 2) in most cases a dose of 100-300 ng/kg/minute must be administered. Norepinephrine will be started on a dose of 100 ng/kg/minute, after which the dosing will be adjusted to achieve the desired blood pressure level. The maximum dose to be used in the study is 1000 ng/kg/minute. Norepinephrine is administered through the central venous catheter.
  Arms: 2

SUMMARY:
The purpose of this study is to test the feasibility of a trial on induced hypertension to improve neurological outcome in patients with subarachnoid haemorrhage that developed the serious complication "delayed cerebral ischemia", and to assess whether induced hypertension results in improved cerebral blood flow (CBF) as measured by means of perfusion-CT.

DETAILED DESCRIPTION:
Background:

Delayed cerebral ischaemia (DCI) is a major complication after aneurysmal subarachnoid haemorrhage (SAH). The proportion of SAH patients who develop DCI is around 30%. Many centres around the world use induced hypertension, alone or in combination with haemodilution and hypervolaemia, so called Triple-H, as standard therapy in the treatment of DCI, but the efficacy of induced hypertension in reducing DCI is based on case series only, and not on a randomised clinical trial.

Objective:

To test the feasibility of a trial on induced hypertension to improve neurological outcome, and to assess whether induced hypertension results in improved cerebral blood flow (CBF) as measured by means of perfusion-CT.

Study design:

A randomised controlled feasibility trial.

Study population:

Patients admitted to the UMC Utrecht after recent SAH, who develop DCI. Twenty four patients will be randomised into a standard care group or one of the intervention groups.

Interventions:

Patients in the intervention groups are treated with induced hypertension (30 mmHg increase in mean arterial pressure) in order to improve CBF. Patients in the standard care group are treated according to the standardised SAH treatment protocol of the UMC Utrecht by monitoring mean arterial pressure and preventing dropping of mean arterial pressure to under 80 mmHg. 24-36 hours after instalment of the treatment, a perfusion CT scan is performed. In patients that do not show any neurological improvement within 24 hours after starting the hypertensive treatment, the administration of norepinephrine will be tapered. In patients who show improvement, induced hypertension will be continued for a total period of 72 hours, after which norepinephrine will be gradually tapered. Measurement of CBF is performed in all participants with perfusion CT-scanning of the brain at the beginning of the study (as part of regular patient care) and after 24-36 hours after starting .

Main outcome measurement:

The number of patients with the diagnosis of DCI after SAH, in which the intervention (induced hypertension) was adequately performed, included within 18 months after the start of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Admission to the UMC Utrecht.
2. Age 18 years or over.
3. Aneurysmal SAH, demonstrated on CT-angiography or cerebral angiography, with onset less than 72 hours before admission.
4. A level of consciousness corresponding to a Glasgow Coma Sum Score above 8, as in patients with lower Glasgow Coma Sum Scores, assessment of further deterioration may be less reliable.

Exclusion Criteria:

1. Symptomatic aneurysm not yet treated by coiling or clipping. Co-existing asymptomatic cerebral aneurysms are no reason for exclusion, since previous studies found no increased risk of rupture of such aneurysms during hypertensive and hypervolemic treatment.(26)
2. Co-existing severe head injury.
3. A history of a cardiac rhythm disorder, necessitating medical treatment.
4. A history of a left ventricular pump failure, necessitating medical treatment.
5. Pregnancy.
6. Known allergy for CT-contrast agents.
7. Renal failure, defined as a serum creatinine > 150 µmol/l, because of the risk of contrast nephropathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-02; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The main study parameter will be the number of SAH patients with a diagnosis of DCI who were randomised to one of the intervention groups, in whom the intervention was adequately performed, during the duration of the trial. | duration of the trial

SECONDARY OUTCOMES:
Related to the inclusion, to the influence on cerebral haemodynamics, to the neurological condition and to adverse events | cerebral haemodynamics: 24-36 hours, neurological condition: 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands